CLINICAL TRIAL: NCT06440343
Title: Effects of Acute Carbohydrate Intake Intra-training in Crosstraining Athletes: a Randomized, Placebo-controlled Crossover Study
Brief Title: Effects of Acute Carbohydrate Intake Intra-training in Crosstraining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Lucas Jurado-Fasoli, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CROSSCARB
Record Dates: First submitted 2024-05-21; First posted 2024-06-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Recovery
Keywords: Sports drink; performance; concurrent exercise; nutrition; recovery
MeSH Terms: interventions — Carbohydrates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carbohydrates (Experimental): 60g of maltodextrin + fructose, 2:1 ratio
  Interventions: Dietary Supplement: Carbohydrates
- Placebo (Placebo Comparator): Preparation of colorants, sweeteners, aromas and acidulants
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Carbohydrates — 60g of maltodextrin + fructose, 2:1 ratio
  Arms: Carbohydrates
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study aims to investigate the effect of acute carbohydrate intake during a crosstraining session on exercise-induced muscle damage and the recovery of crosstraining athletes.

DETAILED DESCRIPTION:
Carbohydrate intake during exercise could decrease the subjective perceived exertion and promote recovery during high-intensity and intermittent exercises such as crosstraining. Nevertheless, despite extensive research on carbohydrate ingestion during exercise across different sports disciplines, its effects have not been investigated in crosstraining sessions.

23 male trained crosstraining athletes will ingest carbohydrates (60g of maltodextrin + fructose, 2:1 ratio) or placebo during a one-and-a-half-hour crosstraining session. The session will consist of a warm-up, a weightlifting part, a strength part, a WOD, and an AMRAP. The rating of perceived exertion (RPE) will be assessed using the validated Borg scale at the beginning of the session, after each part of the training, and at the end of the session. DOMS will be assessed using a visual analog scale at 24 and 48 hours after the crosstraining session.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years.
* Body mass index: 18.5-30 kg/m2.
* Ability to understand the instructions, objectives, and study protocol.
* Minimum of 3 years of experience in crosstraining, with at least 6 hours of weekly training over the past 3 months.
* Resident on the island of Tenerife.

Exclusion Criteria:

* History of a significant adverse cardiovascular event, renal insufficiency, cirrhosis, eating disorder, weight control surgical intervention, or type 2 diabetes mellitus.
* Any chronic condition in which the intake of nutritional supplements is not advisable.
* Any condition that, in the investigator's judgment, would impair the ability to participate in the study or represent a personal risk to the participant.
* Use of medications that may affect the study results.
* Unstable body weight for 3 months prior to the start of the study (> 4 kg loss or gain in - weight).
* Active tobacco abuse or illicit drug use, or history of treatment for alcohol abuse.
* On a special diet or prescribed for other reasons (e.g., celiac disease).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Exercise-induced muscle damage and recovery measured through the countermovement jump | 1 hour 30 minutes
  Countermovement jump height
Exercise-induced muscle damage and recovery through the DOMS scale | 1 hour 30 minutes
  Delayed-onset muscle soreness (DOMS) scale (0-10 arbitrary units)

SECONDARY OUTCOMES:
Capillar lactate levels | 1 hour 30 minutes
  Capillar lactate levels
Capilar glucose levels | 1 hour 30 minutes
  Capilar glucose levels
Subjective fatigue throughe the RPE scale | 1 hour 30 minutes
  Rate of perceived exertion scale
Feeling sensations | 1 hour 30 minutes
  Feeling scale
Performance: Weight used in the crosstraining session | 1 hour 30 minutes
  Weight used in the crosstraining session
Performance: Repetitions performed in the crosstraining session | 1 hour 30 minutes
  Repetitions performed in the crosstraining session
Performance: Rounds performed in the crosstraining session | 1 hour 30 minutes
  Rounds performed in the crosstraining session

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Trivino AR, Diaz-Romero C, Martin-Olmedo JJ, Jimenez-Martinez P, Alix-Fages C, Cwiklinska M, Perez D, Jurado-Fasoli L. Acute effects of intra-training carbohydrate ingestion in CrossFit(R) trained adults: a randomized, triple-blind, placebo-controlled crossover trial. Eur J Appl Physiol. 2025 May;125(5):1337-1347. doi: 10.1007/s00421-024-05689-8. Epub 2024 Dec 13. PMID 39671024